CLINICAL TRIAL: NCT00260234
Title: A Single-Center Phase I/II Study Of Peg-Encapsulated Islet Allografts Implanted In Patients With Type I Diabetes
Brief Title: Safety and Efficacy of PEG-Encapsulated Islet Allografts Implanted in Type I Diabetic Recipients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Stopped in December 2007
Sponsor: Novocell (Industry)
Collaborators: Diabetes & Glandular Disease Research Associates, P.A., San Antonio, TX (Unknown); CHRISTUS Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NC-PCIA-04-001; WIRB #20041068
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Transplantation, Pancreatic Islets; Diabetes Mellitus, Type 1; Insulin Dependent; Islet Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (1):
- PEG Islet Cells (Experimental)
  Interventions: Biological: Allogeneic Cultured Islet Cells (human); Encapsulated

INTERVENTIONS:
Biological: Allogeneic Cultured Islet Cells (human); Encapsulated

SUMMARY:
Insulin dependent Type I diabetics require daily insulin therapy to normalize blood glucose but may have difficulty with significant glycemic excursions and hypoglycemic episodes and crises. Islet cell transplantation can provide relief from daily insulin therapy, normalize blood glucose and reduce or eliminate short and long-term diabetes-related complications. "PEG-Encapsulated Islet Allografts" is a new islet transplant product under development that does not require the ongoing use of immunosuppressive drugs after the implant. This study will test the safety and efficacy of PEG-Encapsulated Islet Allografts in the treatment of Type I diabetes and provide functional outcome measurements.

DETAILED DESCRIPTION:
Allogeneic Cultured Islet Cells (human, Novocell); Encapsulated in Polyethylene Glycol; Administered Subcutaneously are a combination biologic and device product in which the pharmacologically active agent is human insulin that is released from the functional islet cells by natural production and release, stimulated by control mechanisms in response to blood glucose concentrations. The device component is a uniform and conformal polymer coating around each islet. Islet cells are isolated from multiple human pancreases procured from human organ donors who meet a specific human donor profile established by the UNOS and the FDA's requirements for Good Tissue Practices. Because the pancreases used for islet cell isolation are not intended for whole-organ transplantation, specific procurement, surgical removal, packaging and shipping protocols are provided by Novocell, Inc. to the Organ Procurement Organizations.

The primary outcome is demonstration that encapsulated islet allografts can be implanted safely in the subcutaneous tissues without the use of long-term immunosuppression. The expected functional outcomes from the implantation of the encapsulated islets are significant reductions in the average blood glucose daily glycemic excursions and in insulin requirements as well as significant increases in C-peptide levels in response to meal challenges. The ultimate expected outcome is that patients who receive these implants will have reduced hemoglobin A1c levels that may be associated with reduced long-term diabetic complications. An important outcome should be reduction in hypoglycemic episodes and crises with significantly functioning grafts without having the risks associated with hepatic portal vein infusion and long-term immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant non-lactating female subjects > 20 years of age
* Diagnosed with insulin-dependent type I diabetes for at least 20 years
* BMI less than 28 kg/m2
* Insulin requirement less than or equal to 0.7 U/kg/day
* HbA1c greater than or equal to 7.0 %
* Serum C-peptide concentration less than or equal to 0.5 ng/mL stimulated by an OGTT
* Female subjects with childbearing potential must have a negative serum pregnancy test prior to enrollment and must agree to use an effective contraceptive method during the study
* One year of stable diabetes care established in the PI's database without significant changes in insulin requirement or HbA1c or diabetic complication profile

Exclusion Criteria:

* Diagnosis of type II diabetes or maturity onset diabetes of youth (MODY)
* Serum C-peptide greater than 0.5 ng/mL stimulated by OGTT
* Sustained hypertension greater than or equal to 100 mmHg diastolic and/or greater than or equal to 160 mmHg systolic
* History of myocardial infarction or current active cardiac disease
* Current active infection
* Significant renal dysfunction as indicated by GFR less than 80 mL/min/1.73 m2 and/or urinary albumin greater than 500 µg/mL
* Significant liver dysfunction as indicated by ALT or AST more than 3X the upper limit of normal
* Prior whole organ or islet cell transplant
* Concurrent immunosuppressive therapy
* Severe gastroparesis, severe peripheral neuropathy, diabetic foot ulcers, or prior amputations due to diabetic complications
* Any other active autoimmune disease other than autoimmune thyroid disease
* HIV, HBV or HCV positive status
* Uncontrolled or untreated proliferative retinopathy
* Known hypersensitivity or other intolerance to cyclosporine or the inactive ingredients in the product
* Behavioral activities that place the subject at risk in the opinion of the investigator
* Any significant concurrent disease, illness, or psychiatric disorder that would, in the opinion of the investigator, compromise subject safety or compliance, or interfere with consent, study participation, follow-up, or the interpretation of study results
* History of any kind of cancer other than skin cancers (except for melanoma which is exclusionary)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety - will be evaluated by the incidence, grade, and type of adverse events, changes in laboratory parameters, evaluation of the implant site and physical exams.

SECONDARY OUTCOMES:
Efficacy - will be assessed by:
Blood glucose levels
Daily glycemic excursions
Pre-prandial glucose levels
Post-prandial glucose levels
Glucose responses from OGTT (mg/dL and AUC:glucose
Stimulated C-peptide levels from OGTT (ng/mL and
AUC:C-Peptide
HbA1c (%)
Insulin requirements (units/day)
Arginine stimulation tests
Numbers of hypoglycemic and hyperglycemic episodes
Functional duration - will be determined by stimulated C-peptide from OGTT.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwyn Schwartz, M.D., Principal Investigator — Diabetes & Glandular Disease Research Associates, P.A., San Antonio, TX; Paraic Mulgrew, M.D., Principal Investigator — CHRISTUS Santa Rosa Transplant Institute, San Antonio, TX
Locations (2):
- United States (2):
  - CHRISTUS Santa Rosa Transplant Institute, San Antonio, Texas
  - Diabetes & Glandular Disease Research Associates, P.A., San Antonio, Texas

REFERENCES:
- See also: Sponsor's website — http://www.novocell.com
- See also: Diabetes & Glandular Disease Research Associates website — http://www.dgdclinic.com
- See also: CHRISTUS Santa Rosa website — http://www.christussantarosa.org